CLINICAL TRIAL: NCT06711835
Title: Bereitschafts (Readiness) Potential and Reflex Activity During Bone-Loading Exercises
Brief Title: Reflex Activity During Bone-Loading Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eser Kalaoglu (Other Government)
Responsible Party: Sponsor-Investigator, Eser Kalaoglu, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Organization: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IstPRMTRH-EK1
Record Dates: First submitted 2024-11-19; First posted 2024-12-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Reflex; Vibration; Athletic Performance; Bone; Loading exercise

STUDY DESIGN:
Intervention Model Description: This study employs a quasi-experimental design. Participants will be divided into two groups based on their physical activity level: Group 1 (Normally Active Individuals), who engage in typical daily activities without regular sports participation, and Group 2 (Athletic Individuals), who regularly engage in athletic activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Normally Active Individuals) (Experimental): Individuals with Normal Daily Activities
  Interventions: Other: Whole-body vibration and Jumping
- Group 2 (Athletic) (Experimental): Participants who regularly engage in sports activities such as marathon running, basketball, or volleyball
  Interventions: Other: Whole-body vibration and Jumping

INTERVENTIONS:
Other: Whole-body vibration and Jumping — The subjects were first asked to jump in place 20 times, as if they were jumping rope. Then, whole-body vibration was applied. While the participants stood upright on the whole-body vibration device, low-amplitude (1.2 mm) vibrations were applied at eight different frequencies (25, 27, 29, 31, 33, 35, 37, 39 Hz), each lasting for 10 seconds, with a 5-second rest period in between.
  Other Names: Loading exercise

SUMMARY:
Load-bearing exercises are well-established as beneficial for bone health. Their role in promoting healthy bone development and managing osteoporosis is widely recognized. However, the neural mechanisms underlying the positive biomechanical effects of jumping-based load-bearing exercises, such as running, volleyball, basketball, tennis, and skipping rope, remain unclear. The aim of this study is to investigate whether jumping-based load-bearing exercises activate bone myoregulation reflex activity.

DETAILED DESCRIPTION:
Background and Objectives: Wolff was the first to propose that the microarchitectural structure and mechanical resistance of bone are remodeled in response to mechanical loads it experiences. Frost further expanded on this concept with the mechanostat theory, suggesting that bone formation and resorption remain in balance during routine daily activities. Decreased activity leads to increased bone resorption, while increased activity stimulates bone formation. Consequently, the microarchitectural structure and strength of bone weaken or strengthen accordingly. Recently, the bone reflex has been defined, suggesting that the central nervous system controls the local regulatory mechanisms described by Wolff and Frost. The bone reflex describes how osteocytes are stimulated by mechanical loading, leading to the neural regulation of bone formation and resorption according to mechanical needs (bone osteoregulation reflex). Additionally, it describes a mechanism by which the nervous system reflexively regulates the activity of surrounding muscles to optimally position the bone to resist applied mechanical load (bone myoregulation reflex).

Load-bearing exercises are well-established as beneficial for bone health, with their role in promoting healthy bone development and managing osteoporosis being widely recognized. However, the neural mechanisms underlying the positive biomechanical effects of jumping-based load-bearing exercises, such as running, volleyball, basketball, tennis, and rope skipping, remain unclear. The aim of this study is to investigate whether jumping-based load-bearing exercises activate bone myoregulation reflex activity.

Methods: The study will be conducted with a total of 40 healthy volunteers aged 20-50, comprising both women and men. Participants will be recruited from individuals who either regularly engage in jumping-based sports activities (e.g., volleyball, marathon running, and tennis) or those who perform typical daily living activities without regular sports engagement. Participants will be divided into two groups based on their activity levels: Group 1 (Normally Active Individuals) and Group 2 (Athletic Individuals).

Procedures:

Bone myoregulation reflex activity of the soleus and tibialis anterior muscles will be assessed in both groups during whole-body vibration and jumping using surface electromyography.

* Jumping Test: Participants will be instructed to jump in place 20 times, similar to rope skipping, with a 5-second rest interval between each jump.
* Whole-Body Vibration: Participants will stand on the plate and undergo low-amplitude (1.2 mm) whole-body vibration at eight different frequencies (25, 27, 29, 31, 33, 35, 37, and 39 Hz) using a Powerplate Pro5 (Netherlands) device. Each vibration session will last for 10 seconds, with a 5-second rest interval between frequencies.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20-50 years old
* Gender: Male or female
* Health status: Good general health
* Physical activity: Normally Active Individuals or Regularly engaging in jumping sports activities such as volleyball, marathon, or tennis, or not engaging in such activities

Exclusion Criteria:

* Individuals who cannot tolerate whole-body vibration
* Individuals with a history of neuromuscular disease
* Individuals with a history of skeletal disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Bone myoregulation reflex latency | Through study completion, an average of 8 weeks
  The measurement will be taken as the time difference between the moment of mechanical stimulation and the onset of the reflex response in the EMG. The unit of measurement for latency is milliseconds.

SECONDARY OUTCOMES:
Bereitschafts (Readiness) Potential | Through study completion, an average of 8 weeks
  It refers to the myoelectric activity in the tibialis anterior and soleus muscles just before jumping. The onset time of this myoelectric activity will be evaluated in milliseconds, and the amplitude of this activity will be measured in millivolts.

CONTACTS AND LOCATIONS:
Overall Officials: İlhan Karacan, Prof., Study Director — Istanbul Physical Medicine Rehabilitation Training and Research Hospital; Eser Kalaoglu, M.D., Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yildirim MA, Topkara B, Aydin T, Paker N, Soy D, Coskun E, Ones K, Bardak A, Kesiktas N, Ozyurt MG, Celik B, Onder B, Kilic A, Kucuk HC, Karacan I, Turker KS. Exploring the receptor origin of vibration-induced reflexes. Spinal Cord. 2020 Jun;58(6):716-723. doi: 10.1038/s41393-020-0419-5. Epub 2020 Jan 15. PMID 31942042
- [Background] Karacan I, Turker KS. Exploring neuronal mechanisms of osteosarcopenia in older adults. J Physiol. 2026 Jan;604(2):672-688. doi: 10.1113/JP285666. Epub 2024 Aug 9. PMID 39119811
- [Background] Ishikawa S, Kim Y, Kang M, Morgan DW. Effects of weight-bearing exercise on bone health in girls: a meta-analysis. Sports Med. 2013 Sep;43(9):875-92. doi: 10.1007/s40279-013-0060-y. PMID 23754172
- [Background] Zhang L, Miramini S, Richardson M, Ebeling P, Little D, Yang Y, Huang Z. Computational modelling of bone fracture healing under partial weight-bearing exercise. Med Eng Phys. 2017 Apr;42:65-72. doi: 10.1016/j.medengphy.2017.01.025. Epub 2017 Feb 22. PMID 28236603